CLINICAL TRIAL: NCT02544269
Title: Surgical Anesthesia for Elective Hip Surgery - Hemodynamic Effect of Lumbosacral Plexus Blockade Compared to Spinal Anesthesia
Brief Title: Hemodynamic Effect of Lumbosacral Plexus Blockade Versus Spinal Anesthesia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: After pilot study no difference in the primary end point was found between the two primary. Non-inferiority trial not deemed feasible.
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HIP/FUSION#1; 2015-003498-13 (EudraCT Number)
Record Dates: First submitted 2015-09-01; First posted 2015-09-09 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2016-03

CONDITIONS: Total Hip Replacement
Keywords: Lumbosacral plexus blockade; Continuous spinal anesthesia; Hemodynamics
MeSH Terms: interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbosacral plexus blockade (Experimental): Peripheral nerve blockade of lumbar and sacral plexus with ropivacaine max 225 mg perineural
  Interventions: Procedure: Ropivacaine
- Continuous spinal anesthesia (Active Comparator): Continuous spinal anesthesia with plain bupivacaine max 15 mg intrathecal
  Interventions: Procedure: Bupivacaine

INTERVENTIONS:
Procedure: Ropivacaine — Lumbosacral plexus blockade with ropivacaine.
  Arms: Lumbosacral plexus blockade
Procedure: Bupivacaine — Regional anesthesia with bupivacaine titrated to the lowest effective dose
  Arms: Continuous spinal anesthesia

SUMMARY:
The study evaluates the hemodynamic effect of lumbosacral plexus blockades versus spinal anesthesia for hip replacement. Half of participants will receive lumbosacral plexus blockade and the other half will receive continuous spinal anesthesia.

DETAILED DESCRIPTION:
Patients for total hip replacement will be randomized for surgical anesthesia with either lumbosacral plexus blockade or continuous spinal anesthesia. All patients will receive central venous, arterial and spinal catheters. Hemodynamics will be monitored with transpulmonary thermodilution and pulse contour analysis. Perineural injection of study medicine around the lumbar and sacral plexus will be performed guided by ultrasound and nerve stimulation. Study medicine will be injected in divided doses in the spinal catheter. Treatment will be blinded using double-dummy technique. After the first intrathecal dose of study medicine, the hemodynamic response will be monitored for 60 minutes. Patients will then be transferred to the operating room, where total hip replacement will be performed in lumbosacral plexus blockade or spinal anesthesia according to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total hip replacement at Aarhus University Hospital
* Age >= 50 years
* American Society of Anesthesiologists physical status classification score I-III
* Informed consent

Exclusion Criteria:

* Lack of ability to cooperate
* Lack of ability to speak Danish
* Chronic pain, that demands opioid treatment. Not inkl. hip pain.
* Previous venous thromboembolic event
* Previous major back surgery
* Severe cardiopulmonary disease (NYHA class 4)
* Severe untreated hypertension (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 110 mm Hg)
* Obesity (BMI > 35 kg/m^2)
* Pregnancy
* Allergy towards the used local analgetics
* Current treatment with amiodarone or verapamil

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Change of cardiac output | Up to 1 hour
  Change from baseline (before nerve block performance) to 30 minutes after 1st dose of intrathecal study medicine.

SECONDARY OUTCOMES:
Time for performance of nerve blocks | At time of nerve block performance
  Time range (in minutes) from first insertion to last withdrawal of nerve block needle.
Success rate of nerve blocks | 1 day
Change of cardiac stroke volume | Up to 1 hour
  Change from baseline (before nerve block performance) to 30 minutes after 1st dose of intrathecal study medicine.
Change of systemic vascular resistance | Up to 1 hour
  Change from baseline (before nerve block performance) to 30 minutes after 1st dose of intrathecal study medicine.
Change of mean arterial pressure | Up to 1 hour
  Change from baseline (before nerve block performance) to 30 minutes after 1st dose of intrathecal study medicine.
Change of central venous oxygen saturation | Up to 1 hour
  Change from baseline (before nerve block performance) to 30 minutes after 1st dose of intrathecal study medicine.
Maximum plasma concentration of ropivacaine | 80 minutes
  Arterial blood sampling at 20, 40, 60 and 80 minutes after 1st dose of intrathecal study medicine.
Change of plasma concentration of lactate | 60 minutes
  Arterial blood sampling at 0, 30 and 60 minutes after 1st dose of intrathecal study medicine.
Cumulated peroperative propofol dose | Up to 2 hours
Cumulated peroperative opioid dose | Up to 2 hours
Cumulated postoperative opioid dose | Up to 24 hours
Time from end of operation to first opioid dose | Up to 24 hours
Surgeons self reported satisfaction with anesthesia | Up to 2 hours
  Numeric rating scale: 0-10
Patients worst pain during surgery | Up to 2 hours
  Numeric rating scale: 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Niels D Nielsen, MD, Principal Investigator — Aarhus University, Dept. of Clinical Medicine; Thomas F Bendtsen, MD, PhD, Study Director — Aarhus University Hospital, Dept. of Anesthesiology
Locations (1):
- Center for Planlagt Kirurgi, Silkeborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be made available through Danish Data Archive.